CLINICAL TRIAL: NCT06452212
Title: A Non-Interventional, Modified Delphi Study to Establish Consensus Recommendations on the Optimal Management of Metastatic Hormone-Sensitive Prostate Cancer (mHSPC) Patients in South Korea
Brief Title: Non-Interventional Study to Establish Consensus on Management of Metastatic Hormone-Sensitive Prostate Cancer Patients
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 9785-MA-3541
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Hormone-Sensitive Prostate Cancer
Keywords: mHSPC; Urological cancers
MeSH Terms: conditions — Urologic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Urologists: Health care professionals/panelist.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No investigational drug will be administered to participants in this study.

SUMMARY:
The purpose of this study is to establish an expert consensus recommendations on managing patients with mHSPC in South Korea, and to provide clinicians with a comprehensive guide to support their clinical decision making. There are no secondary objectives for this study.

DETAILED DESCRIPTION:
Data collection for this study will be conducted through 2 rounds of web-based surveys of health care professionals (HCPs). A meeting with the panelists will be held as a 3rd round if a consensus for pre determined key questions is not achieved after the 2 rounds of the survey.

ELIGIBILITY:
Inclusion Criteria:

* Urologist from university hospitals in South Korea.
* Has a minimum 10 years of practice experience (experience as a military or public health doctor could be considered practice experience)
* Sees a minimum of 50 mHSPC patients in a year.
* At least 10 publications in SCIE (Science Citation Index Expanded) journals in the past 5 years.

Exclusion Criteria:

* Urologist in private practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target recruitment of 25 urologists will be recruited with an acceptable goal of 20 as panelists from university hospitals in South Korea.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Treatment plans for patients with mHSPC | Up to 7 days
  Treatment plans for patients with mHSPC within the local healthcare environment will be collected via online surveys and a consensus meeting will be held if required.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Korea, Inc.
Locations (1):
- KR82001, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.